CLINICAL TRIAL: NCT02016976
Title: Effect of Local Anesthetic EMLA (Lidocaine 2.5% and Prilocaine 2.5%) Cream and Reduction in Dose, Pain and Intravenous Analgesic During Permanent Pacemaker Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0094-13-HYMC
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Pacemaker Implantation; Pain
MeSH Terms: conditions — Pain | interventions — Midazolam; Meperidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMLA analgesic cream (Active Comparator): Patients who have had EMLA analgesic cream applied to area before pacemaker implantation
  Interventions: Drug: EMLA Analgesic Cream
- Routine treatment (Active Comparator): Patients who have received routine treatment (Dormicum 2.5 mg and Pethidine 25 mg) before and during pacemaker implantation
  Interventions: Drug: Dormicum 2.5 mg and Pethidine 25 mg

INTERVENTIONS:
Drug: EMLA Analgesic Cream
  Arms: EMLA analgesic cream
Drug: Dormicum 2.5 mg and Pethidine 25 mg — Routine anesthesia and analgesia ( Dormicum 2.5 mg and Pethidine 25 mg )normally given to patients before and during pacemaker implantation
  Arms: Routine treatment

SUMMARY:
The investigators believe that the local anesthetic EMLA (Lidocaine 2.5% and Prilocaine 2.5%) cream will lessen pain and reduce the need for anesthesia and analgesia, when implanting a permanent pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing pacemaker implantation

Exclusion Criteria:

* Dementia Patients
* Psychiatric Patients
* Unconscious Patients
* Patients with sensitivity to EMLA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | One hour
  EMLA anesthetic cream will be applied to area where pacemaker is to be implanted. Pain reduction will be measured using the visual analog scale (VAS) at three intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel